CLINICAL TRIAL: NCT06908837
Title: Effects of 10 Versus 20 mL Local Anesthetic for Popliteal Plexus Block on Opioid Consumption, Pain, and Patient-Reported Outcomes After Total Knee Arthroplasty - a Randomized, Controlled, Blinded Study
Brief Title: Effects of 10 Versus 20 mL Local Anesthetic for Popliteal Plexus Block on Opioid Consumption, Pain, and Patient-Reported Outcomes After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Responsible Party: Principal Investigator, Johan Kløvgaard Sørensen, Principal Investigator, Regionshospitalet Silkeborg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-520204-26-00
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Arthroplasty; Regional Anesthesia; Multimodal Analgesic Approach; Postoperative Opioid-related Complications
Keywords: Popliteal Plexus Block; Total knee arthroplasty; regional anesthesia; optimal analgesic volume; postoperative pain; postoperative opioid consumption; Quality of Recovery 15; Manual Muscle Test; Postoperative mobility
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This single-centre, blinded, controlled, randomized clinical trial follows a parallel design, with one group receiving a PPB with 10 mL of bupivacaine 5 mg/mL and the other group receiving a PPB with 20 mL of bupivacaine 5 mg/mL. A total of 120 patients will be included and allocated in a 1:1 ratio using computer-generated block randomization (blocks of 10).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Good-Clinical-Practice monitor is also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Popliteal Plexus Block with 20 mL of bupivacaine (Experimental)
  Interventions: Drug: Bupivacaine
- Popliteal Plexus Block with 10 mL of bupivacaine (Active Comparator)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Applied perineurally using a 22-gauge, 80-mm block needle (Temena, Felsberg, Germany) under ultrasound guidance.

SUMMARY:
This trial aims to assess the analgesic effect of Popliteal Plexus Block (PPB) with 10 mL versus 20 mL of Bupivacain 5 mg/mL, when applied as an adjunct treatment to a multimodal analgesic regimen following primary total knee arthroplasty. We hypothesize that PPB with 20 mL of local anesthetic reduces 24-hour postoperative opioid consumption (= primary outcome) compared to 10 mL after TKA.

Secondary outcome include

* the frequency of 24-hour opioid-free analgesia
* pain intensity at rest and during mobilization
* Manual Muscle Tests and ability to mobilize with crutches six hours after end-of-surgery
* and patients reported outcomes using the Quality of Recovery 15 survey 24 hours after end-of-surgery.

Participant will:

* undergo primary total knee arthroplasty in spinal anesthesia.
* recieve a PPB with either 10 mL of Bupivacaine or 20 mL.
* recieve a multimodal analgesic regime including a Femoral Triangle Block.
* Have 10 scored morphine tablets available for self-administration within the first 24 postoperative hours after end-of-surgery.
* be examined by a physiotherapist 6 hours (±1 hour) after end-of-surgery to assess pain scores, manual muscle testing of ankle and knee function, and the ability to mobilize with crutches.
* complete a survey 24 hours after end-of-surgery to assess self-administered morphine intake, pain scores, and Quality of Recovery-15.

DETAILED DESCRIPTION:
Patients will undergo primary unilateral total knee arthroplasty with insertion of non-cruciate retaining standard cemented prosthesis by a parapatellar medial approach, without use of tourniquet or Local Infiltration Analgesia.

For the spinal anesthesia, 3 mL of Ropivacaine 5 mg/ml will be applied.

All patients will receive a femoral triangle block in combination with the PPB, both administered immediately after surgery in the post-anesthesia care unit.

Description of the PPB procedure:

The superficial femoral artery is identified at mid-thigh level and traced caudally until it deviates from sartorius muscle and is positioned adjacent to the posteromedial margin of the vastus medialis muscle, close to the adductor hiatus. The needle will be inserted medially to the transducer and advanced in-plane through the sartorius muscle targeting the endpoint of injection in the distal part of the adductor canal, on the top of the superficial femoral artery, posteromedial to the fascia of the vastus medialis muscle. We will inject the allocated volume of bupivacaine 5 mg/mL, ensuring anterolaterally spread to the artery

The Femoral Triangle Block uses 15 mL of Bupivacaine 5 mg/mL (10 mL applied in the femoral triangle to target the saphenous nerve and nerve to vastus medialis and 5 mL applied to target the intermediate femoral cutaneous nerve located at the superficial side of the sartorius muscle).

The multimodal analgesic regime also consists of a Dexamethasone 12 mg IV (administered perioperatively), Paracetamol (1000 mg) x 4 daily + NSAID (400 mg) x 3 times daily postoperatively, inclusing preoperatively administration of Paracetamol 1000 mg and Ibuprofen 400 mg.

The scored morphine tablets allows the patients to take 5 mg morphine at a time, with a maximum oral dose of 100 mg within the first 24 hours after end-of-surgery time. If needed, hospital staff can administer rescue doses of intravenous morphine, which will be recorded in the patient file. Total opioid consumption will be reported as oral morphine milligram equivalents (MME), combining hospital-administered opioid doses from the patient file and self-reported intake of dispensed morphine tablets.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary total knee arthroplasty in spinal anesthesia.
* Ability to give their written informed consent after having fully understood the contents of the study.
* American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.

Exclusion Criteria:

* Patients who cannot read or speak Danish.
* Patients who cannot operate or have access to a smartphone with internet connectivity (required for patient-reported outcome assessment).
* Patients with allergies or intolerance to the medicines used in the study.
* Patients with a consistent daily intake of opioids preoperatively.
* Patients who are dependent on walking aid devices preoperatively.
* Patients suffering from alcohol and/or drug abuse - based on the investigator's assessment.
* BMI > 40.
* Diagnosed with chronic neurodegenerative disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption, expressed in oral morphine milligram equivalents (MME). | From T0 (end-of-surgery time) to T24 (24 hours after end-of-surgery time)
  Combining hospital-administered opioid doses from the patient file and self-reported intake of dispensed morphine tablets.

SECONDARY OUTCOMES:
No opioid requirement | From T0 (end-of-surgery time) to T24 (24 hours after end-of-surgery time)
  The frequency of patients with no opioid consumption
Pain at rest | Assessed preoperatively, at T6 (6±1 hours after end-of-surgery time), and at T24 (24 hours after end-of-surgery time).
  Registered using the Numeric Rating Scale (0 = no pain and 10 = worst imaginable pain)
Pain during 10 meters walk assisted only by crutches | Assessed preoperatively, at T6 (6±1 hours after end-of-surgery time), and at T24 (24 hours after end-of-surgery time).
  Registered using the Numeric Rating Scale (0 = no pain and 10 = worst imaginable pain)
Early postoperative walking ability | Assessed at T6 (6±1 end-of-surgery time)
  The frequency of patients unable to walk 10 meters with crutches at T6
Postoperative Manual Muscle Test | Assessed at T6 (6±1 end-of-surgery time)
  Frequency of patients with Manual Muscle Test results < Grade 3 in evaluations of dorsiflexion and plantarflexion of the ankle and knee extension.
  Grade 5: Patient can move the limb in the intended direction against gravity and maximum manual resistance. Grade 4: Patient can move the limb in the intended direction against gravity and moderate manual resistance. Grade 3: Patient can move the limb in the intended direction against gravity without resistance. Grade 2: Patient can move the limb in the intended direction only by elimination of the gravity or with minimal assistance from the investigator. Grade 1: Patient is unable to move the limb in the intended direction, but muscle contraction of the respective muscle is palpable or observable. Grade 0: No muscle contraction of the respective muscle is palpable or observable.
Quality of Recovery 15 | Assessed at T24 (24 hours after end-of-surgery time)
  Patient reported outcome measure of the Quality of Recovery 15 survey.

CONTACTS AND LOCATIONS:
Overall Officials: Johan K Sørensen, MD, Principal Investigator — Elective Surgery Centre at Silkeborg Regional Hospital, Denmark
Locations (1):
- Elective Surgery Centre at Silkeborg Regional Hospital, Silkeborg, Denmark Central Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data is available upon reasonable request.

REFERENCES:
- [Derived] Sorensen JK, Jensen MSH, Grevstad U, Nikolajsen L, Runge C. Optimal Analgesic Volume for Popliteal Plexus Block After Total Knee Arthroplasty: A Blinded RCT Protocol. Acta Anaesthesiol Scand. 2025 Jul;69(6):e70057. doi: 10.1111/aas.70057. PMID 40346895